CLINICAL TRIAL: NCT05856539
Title: Erector Spinae Plane Block in Patients Undergoing Minimally Invasive Lumbar Spine Surgery: A Randomized Controlled Trial
Brief Title: ESP Block in MIS Lumbar Spine Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-1386
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Patients With Spinal Stenosis Indicated for MIS TLIF
Keywords: Erector spinae plane (ESP) block; Transforaminal lumbar interbody fusion (TLIF); Minimally invasive spine surgery; Lumbar spine; Spinal fusion
MeSH Terms: conditions — Bites and Stings | interventions — Parapsychology; Dental Occlusion

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, randomized controlled trial.
Who Masked: Participant
Masking Description: Patients will be blinded to randomization (whether or not they received an ESP block preoperatively). Co-investigators will not be blinded as the anesthesiologist will need to perform the ESP block.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ESP Block (Experimental): Patients assigned to the "ESP Block" arm will receive an ESP block prior to the surgery.
  Interventions: Procedure: Erector spinae plane (ESP) block
- Control (No Intervention): Patients assigned to the "Control" group will not receive an ESP block prior to the surgery.

INTERVENTIONS:
Procedure: Erector spinae plane (ESP) block — ESP block is an opioid-sparing regional anesthetic involving bupivacaine and dexamethasone for lumbar spinal surgery with touted benefits including opioid use reduction and improved pain control.
  Arms: ESP Block

SUMMARY:
This is a prospective, randomized controlled trial of patients undergoing minimally invasive transforaminal lumbar interbody fusion. This study will randomize patients into one of two groups: erector spinae plane (ESP) block and no ESP block.

DETAILED DESCRIPTION:
Minimally invasive (MIS) spinal surgical procedures such as MIS transforaminal lumbar interbody fusion (TLIF) are being increasingly performed due to reduced morbidity. However, the mainstay for perioperative analgesia after these surgeries remains to be opioid pain medications, which have a number of associated adverse effects such as respiratory depression, hyperalgesia, and opioid habituation. Recently, the erector spinae plane (ESP) block has been introduced as an opioid-sparing regional anesthetic for lumbar spinal surgery with touted benefits including opioid use reduction and improved pain control. The proposed study aims to enroll patients in a double blind randomized controlled trial to undergo MIS TLIF with an ESP block or as conventional control group. Preoperative patient demographics, comorbidities, history of opioid use, and operative details will be obtained. Comprehensive assessment of opioid utilization, postoperative pain, non-opioid pain medication use, opioid-induced complications, time to opioid cessation, time to physical therapy clearance, length of stay, as well as other related outcomes will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Patients scheduled for MIS TLIF (any level) with the principal investigator
* ASA 1, 2, 3

Exclusion Criteria:

* ASA 4 or higher
* BMI >40
* Chronic opioid use (daily use for > 3 months)
* Revision surgery, any history of previous lumbar spine surgery
* Allergy to any of the study medications
* Non-English speaking
* Chronic renal insufficiency or failure (creatinine >2) or severe hepatic disease (cirrhosis, failure)
* Pregnancy
* Any concomitant surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
24-hour oral morphine milligram equivalents (OMEs) | 24 hours postoperatively
  The primary outcome of the study will be cumulative opioid use in the first 24 hours postoperatively in oral morphine milligram equivalents (OMEs) (24 hour period from PACU admission to POD1).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Only the PI, study coordinators listed on the IRB protocol, and co-investigators will have access to the IPD information.

REFERENCES:
- [Background] De Rojas JO, Syre P, Welch WC. Regional anesthesia versus general anesthesia for surgery on the lumbar spine: a review of the modern literature. Clin Neurol Neurosurg. 2014 Apr;119:39-43. doi: 10.1016/j.clineuro.2014.01.016. Epub 2014 Jan 27. PMID 24635923
- [Background] Dunn LK, Durieux ME, Nemergut EC. Non-opioid analgesics: Novel approaches to perioperative analgesia for major spine surgery. Best Pract Res Clin Anaesthesiol. 2016 Mar;30(1):79-89. doi: 10.1016/j.bpa.2015.11.002. Epub 2015 Nov 24. PMID 27036605
- [Background] Garcia RM, Cassinelli EH, Messerschmitt PJ, Furey CG, Bohlman HH. A multimodal approach for postoperative pain management after lumbar decompression surgery: a prospective, randomized study. J Spinal Disord Tech. 2013 Aug;26(6):291-7. doi: 10.1097/BSD.0b013e318246b0a6. PMID 23887076
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Tulgar S, Kapakli MS, Senturk O, Selvi O, Serifsoy TE, Ozer Z. Evaluation of ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy: A prospective, randomized, controlled clinical trial. J Clin Anesth. 2018 Sep;49:101-106. doi: 10.1016/j.jclinane.2018.06.019. Epub 2018 Jun 15. PMID 29913392
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH, Kilic CT. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. J Clin Anesth. 2018 Nov;50:65-68. doi: 10.1016/j.jclinane.2018.06.033. Epub 2018 Jul 2. PMID 29980005
- [Background] Krishna SN, Chauhan S, Bhoi D, Kaushal B, Hasija S, Sangdup T, Bisoi AK. Bilateral Erector Spinae Plane Block for Acute Post-Surgical Pain in Adult Cardiac Surgical Patients: A Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2019 Feb;33(2):368-375. doi: 10.1053/j.jvca.2018.05.050. Epub 2018 Jun 4. PMID 30055991
- [Background] Abu Elyazed MM, Mostafa SF, Abdelghany MS, Eid GM. Ultrasound-Guided Erector Spinae Plane Block in Patients Undergoing Open Epigastric Hernia Repair: A Prospective Randomized Controlled Study. Anesth Analg. 2019 Jul;129(1):235-240. doi: 10.1213/ANE.0000000000004071. PMID 30801359
- [Background] Yang HM, Choi YJ, Kwon HJ, O J, Cho TH, Kim SH. Comparison of injectate spread and nerve involvement between retrolaminar and erector spinae plane blocks in the thoracic region: a cadaveric study. Anaesthesia. 2018 Oct;73(10):1244-1250. doi: 10.1111/anae.14408. Epub 2018 Aug 16. PMID 30113699
- [Background] Adhikary SD, Bernard S, Lopez H, Chin KJ. Erector Spinae Plane Block Versus Retrolaminar Block: A Magnetic Resonance Imaging and Anatomical Study. Reg Anesth Pain Med. 2018 Oct;43(7):756-762. doi: 10.1097/AAP.0000000000000798. PMID 29794943
- [Background] Melvin JP, Schrot RJ, Chu GM, Chin KJ. Low thoracic erector spinae plane block for perioperative analgesia in lumbosacral spine surgery: a case series. Can J Anaesth. 2018 Sep;65(9):1057-1065. doi: 10.1007/s12630-018-1145-8. Epub 2018 Apr 27. PMID 29704223
- [Background] Cesur S, Yayik AM, Ozturk F, Ahiskalioglu A. Ultrasound-guided Low Thoracic Erector Spinae Plane Block for Effective Postoperative Analgesia after Lumbar Surgery: Report of Five Cases. Cureus. 2018 Nov 16;10(11):e3603. doi: 10.7759/cureus.3603. PMID 30680264
- [Background] Ueshima H, Inagaki M, Toyone T, Otake H. Efficacy of the Erector Spinae Plane Block for Lumbar Spinal Surgery: A Retrospective Study. Asian Spine J. 2019 Apr;13(2):254-257. doi: 10.31616/asj.2018.0114. Epub 2018 Nov 15. PMID 30424594
- [Background] Singh S, Chaudhary NK. Bilateral Ultasound Guided Erector Spinae Plane Block for Postoperative Pain Management in Lumbar Spine Surgery: A Case Series. J Neurosurg Anesthesiol. 2019 Jul;31(3):354. doi: 10.1097/ANA.0000000000000518. No abstract available. PMID 29965831
- [Background] Singh S, Choudhary NK, Lalin D, Verma VK. Bilateral Ultrasound-guided Erector Spinae Plane Block for Postoperative Analgesia in Lumbar Spine Surgery: A Randomized Control Trial. J Neurosurg Anesthesiol. 2020 Oct;32(4):330-334. doi: 10.1097/ANA.0000000000000603. PMID 31033625
- [Background] Yayik AM, Cesur S, Ozturk F, Ahiskalioglu A, Ay AN, Celik EC, Karaavci NC. Postoperative Analgesic Efficacy of the Ultrasound-Guided Erector Spinae Plane Block in Patients Undergoing Lumbar Spinal Decompression Surgery: A Randomized Controlled Study. World Neurosurg. 2019 Jun;126:e779-e785. doi: 10.1016/j.wneu.2019.02.149. Epub 2019 Mar 8. PMID 30853517